CLINICAL TRIAL: NCT05890287
Title: An Open, Single-center, Exploratory Cohort Study of Chidamide in Combination With Endocrine in Maintenance Therapy After First-line Chemotherapy for HR+/HER2- Breast Cancer
Brief Title: A Study of Chidamide Plus Endocrine in Maintenance Treatment of HR+/HER2- Breast Cancer After First-line Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Li Zhang, Deputy chief physician, Tianjin Medical University Cancer Institute and Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C44
Record Dates: First submitted 2023-05-11; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: HR Positive HER2 Negative Advanced Breast Cancer
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; exemestane; Fulvestrant; Letrozole; Anastrozole; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A in advanced stages of first-line ± endocrine therapy without CDK4/6 inhibitors (Experimental): Chidamide tablets, specification 5mg/ tablet. Administration method: Oral, 30mg/ time, twice a week; Endocrine drugs: (TAM, AI, fluvestran, etc.) According to patients' previous endocrine treatment, different endocrine drugs were selected according to researchers' judgment, and the dosage was used according to the instructions; OFS drugs (for premenopausal patients only).
  Interventions: Drug: Chidamide
- Late-stage first-line ± endocrine therapy with CDK4/6 inhibitors in cohort B (Experimental): Chidamide tablets, specification 5mg/ tablet. Administration method: Oral, 30mg/ time, twice a week; Endocrine drugs: (TAM, AI, fluvestran, etc.) According to patients' previous endocrine treatment, different endocrine drugs were selected according to researchers' judgment, and the dosage was used according to the instructions; OFS drugs (for premenopausal patients only).
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide+ exemestane/Fulvestrant/Letrozole/Anastrozole/Tamoxifen
  Other Names: exemestane; Fulvestrant; Letrozole; Anastrozole; Tamoxifen

SUMMARY:
To explore the efficacy and safety of Chidamide combined with endocrine for maintenance therapy after first-line chemotherapy for HR+/HER2- breast cancer

DETAILED DESCRIPTION:
o explore the efficacy and safety of Chidamide combined with endocrine drug maintenance after first-line chemotherapy in the treatment of advanced untreated breast cancer; To explore the efficacy and safety of Chidamidecombined with endocrine drugs after first-line chemotherapy in the treatment of advanced first-line non-chemotherapeutic breast cancer after failure of CDK4/6 inhibitors

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal/premenopausal women aged ≥18 years and ≤70 years;
2. HR + / HER2 breast cancer confirmed by histology (note: her2-negative is defined as: (1) IHC1 + / IHC0; ②IHC2+ : FISH-);
3. Confirmed by the histology of locally advanced breast cancer (local treatment) to radical or recurrent metastatic breast cancer;
4. In the late stage of untreated or experienced a CDK4/6 with endocrine therapy of patients;
5. Researchers think that for selecting patients with chemotherapy (step 2022 guidelines recommend for internal transfer, always endocrine therapy resistance or preferred to rescue patients with endocrine therapy best choice of chemotherapy);
6. One line finish cycle disease after chemotherapy (4 to 8 cycles) to alleviate or stable, quasi follow-up maintenance treatment: a. late stage A gleam of unused CDK4/6 inhibitors + endocrine group subjects into the queue for A; b. Used in the late phase line CDK4/6 inhibitors queue B + endocrine subjects into groups;
7. Into the former group at least one measurable lesions (RECIST v1.1 standard); 8.ECOG score 0 to 2 points;

9.Always all the acute toxic reaction caused by antineoplastic therapy in screening before easing to 0 and 1 level (according to the NCI CTCAE 5.0 judgment; Hair loss, other than toxicity that the investigator believes does not pose a safety risk to the subject); 10. Functions: bone marrow neutrophils absolute acuity 1.5 x 109 / L, platelet acuity 100 x 109 / L, 90 g/L or higher hemoglobin; 11. Liver and kidney function: TBIL acuities were 1.5 x ULN; ALT and AST≤2.5 x ULN; In case of liver metastasis, ALT and AST≤ 5×ULN; BUN and Cr≤1.5×ULN and creatinine clearance ≥50 ml/min; 12.Voluntary participation in the clinical trials, signed written informed consent.

Exclusion Criteria:

1. Factors that significantly affect oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
2. Always received HDACi anti-tumor treatment;
3. This scheme known drug components have allergy history;
4. Always with other malignant tumours within five years, not including has cured thyroid papillary carcinoma, cervical carcinoma in situ, basal cell carcinoma or skin squamous cell carcinoma of the skin;
5. Within 4 weeks before into the group participated in other clinical trials;
6. A history of immune deficiency, including test positive for HIV, or has other acquired, congenital immunodeficiency disease, or has a history of organ transplantation;
7. Unable to control the important cardiovascular disease: a history of clinical significance of long QT, stage or screen between QTc > 450 ms; Severe cardiovascular injury (greater than a New York Heart Association (NYHA) Class II history of congestive heart failure), unstable angina or myocardial infarction within the last 6 months, or severe arrhythmia;
8. Pregnancy and lactation women patients or in infertile women baseline pregnancy test positive; Or participants of childbearing age who were unwilling to use effective contraception during the study period and for at least 8 weeks after the last dosing;
9. According to the researcher's judgment, there is serious to endanger the safety of patients, the patients completed studies or associated with disease (such as severe hypertension, diabetes, thyroid disease, active infection, etc.);
10. Always have a clear history of neurological or psychiatric disorders, including epilepsy or dementia, etc.;
11. Reference: subjects had active hepatitis (hepatitis b positive HBsAg and HBV DNA of 500 IU/ml or more; Hepatitis C reference: HCV antibody positive and HCV virus copy number > upper limit of normal);
12. The researchers determine doesn't fit to the researchers.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 year
  PFS is defined as the time from the date of treatment to the first date of disease

SECONDARY OUTCOMES:
Objective response rate | 2 year
  Treatment response are defined as complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) according to Response Evaluation Criteria in Solid Tumor (RECISIT criteria, version 1.1). The percentage of patients who achieved CR and PR was defined as objective response rate (ORR)
Disease control rate | 2 year
  his means that in all patients with a tumor who receive a certain treatment, the tumor shrinks or stays stable, and stays that way for a certain amount of time
Clinical Benefit Rate (CBR) | 2 year
  CBR is defined as the rate of patients who achieved complete response, partial response, and stable disease for >= 24 weeks as the best response of treatment.
Overall Survival (OS) | 2 year
  OS defined as the time from the first study treatment administration to death from any cause
Adverse events (AE) | 2 year
  The level of the adverse event (AE) is analyzed according to the Common Terminology Criteria for Adverse Event (CTCAE) (version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- 天津市肿瘤医院, Tianjin, China

IPD SHARING:
Plan to Share IPD: No